CLINICAL TRIAL: NCT01684917
Title: Application of New Technologies and Tools to Nutrition Research
Acronym: NutriTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: 12/L0/0139
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; Metabolites
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Life style advice (Experimental): reduce energy intake by 20% less than estimated energy expenditure.
  Interventions: Behavioral: Metabolomic and Energy Intake Restriction
- UK background diet (Active Comparator): Diet where energy intake will be matched with estimated energy expenditure.
  Interventions: Behavioral: Metabolomic and Energy Intake Restriction
- Metabolomic inquiry (Other): This inquiry took place prior to the randomized controlled trial and include 50 volunteers who will then be asked to volunteers of the weight loss study. Were randomly assigned to one of five different diets; red meat, fish, poultry, processed meat or a supplement and vegetarian option.
  Interventions: Behavioral: Metabolomic and Energy Intake Restriction

INTERVENTIONS:
Behavioral: Metabolomic and Energy Intake Restriction — Metabolomic inquiry followed by a 12 week energy intake restriction. This study is part of a very large European study called EPIC. Only the results by Lee et al. 2016 have been presented here. The results of the study published by Cheung 2017 are from a different study. therefore the entries for the results are correct. For this particular study, participants were not randomly assigned to one of five different diets; red meat, fish, poultry, processed meat or a supplement and vegetarian option. In summary, both studies (lee and cheung) are considered as separate trials and results of the first phase where participants were assigned to one of five different diets, are reported separately. Unfortunately no different NCT number is available.
  Other Names: Energy restriction diet; Metabolomic

SUMMARY:
The overall objective of the research is to develop new methods for studying the link between diet, health and disease.

DETAILED DESCRIPTION:
The enquiry consists of two part. A metabolomic biomarker discovery study followed by a randomised controlled trial of moderate dietary induced weight loss.

A cohort of moderately overweight men and women will undergo a metabolomic study follow by randomised controlled trial of a healthy diet with a 20% energy restriction for a 12 week period. This intervention will improve the volunteer's body composition and reduce their risk of developing diabetes.

Extensive tests will be conducted before and after the dietary intervention using emerging technologies with current state-of-the-art methods. These tests will monitor the numerous physiological adaptations that have occurred on a gene, cell, organ and organismic level.

The study will, therefore, aim for a scientific breakthrough by developing a series of novel biological "markers" that can accurately determine an individual's health status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight volunteers (body mass index (BMI) of 25-30 kg/m2)
* Age between 50-65 years

Exclusion Criteria:

* Weight change of ≥ 3kg in the preceding 3 months
* Current smokers
* Substance abuse
* Excess alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Have any metallic or magnetic implants such as pacemakers
* Use of medications likely to interfere with energy metabolism, appetite regulation and hormonal balance, including: anti inflammatory drugs or steroids, antibiotics, androgens, phenytoin, erythromycin or thyroid hormones.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Frost, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Result] Lee S, Norheim F, Langleite TM, Noreng HJ, Storas TH, Afman LA, Frost G, Bell JD, Thomas EL, Kolnes KJ, Tangen DS, Stadheim HK, Gilfillan GD, Gulseth HL, Birkeland KI, Jensen J, Drevon CA, Holen T; NutriTech Consortium. Effect of energy restriction and physical exercise intervention on phenotypic flexibility as examined by transcriptomics analyses of mRNA from adipose tissue and whole body magnetic resonance imaging. Physiol Rep. 2016 Nov;4(21):e13019. doi: 10.14814/phy2.13019. PMID 27821717
- [Result] Cheung W, Keski-Rahkonen P, Assi N, Ferrari P, Freisling H, Rinaldi S, Slimani N, Zamora-Ros R, Rundle M, Frost G, Gibbons H, Carr E, Brennan L, Cross AJ, Pala V, Panico S, Sacerdote C, Palli D, Tumino R, Kuhn T, Kaaks R, Boeing H, Floegel A, Mancini F, Boutron-Ruault MC, Baglietto L, Trichopoulou A, Naska A, Orfanos P, Scalbert A. A metabolomic study of biomarkers of meat and fish intake. Am J Clin Nutr. 2017 Mar;105(3):600-608. doi: 10.3945/ajcn.116.146639. Epub 2017 Jan 25. PMID 28122782
- [Derived] Donado-Pestana CM, Rodrigues L, Rundle M, Thomas EL, Wopereis S, Gundersen TE, Trezzi JP, Bunzel D, Kiselova-Kaneva Y, Sonntag D, Kulling SE, Ivanova D, Hiller K, Drevon CA, Brennan L, Bell JD, van Ommen B, Frost G, Daniel H, Fiamoncini J. Plasma metabolomic profiles reveal sex-specific response to an oral glucose tolerance test in late middle-aged adults. Mech Ageing Dev. 2025 Aug;226:112081. doi: 10.1016/j.mad.2025.112081. Epub 2025 Jun 2. PMID 40467008
- [Derived] Yin X, Gibbons H, Rundle M, Frost G, McNulty BA, Nugent AP, Walton J, Flynn A, Gibney MJ, Brennan L. Estimation of Chicken Intake by Adults Using Metabolomics-Derived Markers. J Nutr. 2017 Oct 1;147(10):1850-1857. doi: 10.3945/jn.117.252197. PMID 28794208

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: An overweight/dysglycemic group
  4 h of intense exercise each week, including two whole-body strength-training sessions and two spinning bike interval sessions for 12 weeks
- Diet: overweight/ obese subjects with normal glucose metabolism with energy restriction, 20% reduced intake of energy from food for 12 weeks.
  Energy intake was matched with estimated energy expenditure
- Exercise, Control: An overweight with no dysglycemia 4 h of intense exercise each week, including two whole-body strength-training sessions and two spinning bike interval sessions for 12 weeks
- Diet, Control: overweight/ obese subjects with normal glucose metabolism for 12 weeks
  Energy intake was matched with estimated energy expenditure
Period: Overall Study
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Started | 11 | 7 | 13 | 5
Completed | 11 | 7 | 13 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diet: overweight/ obese subjects with normal glucose metabolism with energy restriction, 20% reduced intake of energy from food for 12 weeks
- Diet, Control: overweight/ obese subjects with normal glucose metabolism for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control | Total
Number analyzed (Participants) | 11 | 7 | 13 | 5 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (1.7) | 59 (1.3) | 50 (2.1) | 57 (2.7) | 55 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 2 | 6
  Male | 11 | 3 | 13 | 3 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 7 | 13 | 5 | 36
BMI [Mean (Standard Deviation); unit: kg/m^2] — As shown in table 1 of the publication by Lee at al 2016, the unit measure used was kg/m2.
  kg/m^2 | 28.9 (2.5) | 30.8 (3.1) | 23.5 (2) | 29.1 (2) | 28 (2.3)
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] — As shown in table 1 of the publication by Lee at al 2016, the unit measure used was mmol/L.
  mmol/L | 5.8 (0.4) | 5.0 (0.6) | 5.4 (0.1) | 4.6 (0.3) | 5.2 (0.4)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] — As shown in table 1 of the publication (Lee et al 2016), the unit measure for cholesterol is mg/dL.
  mg/dL | 5.6 (0.5) | 5.6 (1.2) | 5.1 (0.2) | 4.9 (0.3) | 5.2 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Glucose Infusion rate assessed by the euglycemic hyperinsulinemic clamp. Insulin Sensitivity assessment was only performed in the "Exercise" and "Exercise, Control" groups. No data were collected for this Outcome from the remaining groups.
Time Frame: Baseline, 12 weeks
Population: No data available for diet and diet-control group
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 11 | 0 | 13 | 0
mg/kg/min
  Baseline | 4.2 (1.8) |  | 7.6 (1.6) |
  12 weeks | 5.4 (1.8) |  | 10.4 (2.6) |
Statistical Analysis 1: Comparison: Exercise; Baseline vs 12 weeks; Test type: Superiority; p < 0.05, t-test, 2 sided — calculated. The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance
Statistical Analysis 2: Comparison: Exercise, Control; Baseline vs 12 weeks; Test type: Superiority; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Metabolomic Biomarker Discovery - Changes in Blood Plasma Cholesterol
Description: Changes in blood plasma cholesterol in mg/dL- baseline to 12 weeks, after treatment. Statistical Analysis was performed only for the "Diet" Arm/Group.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 11 | 7 | 13 | 5
mg/dL
  Baseline | 5.6 (0.5) | 5.6 (1.2) | 5.1 (0.2) | 4.9 (0.3)
  12 weeks | 5.8 (0.7) | 4.9 (1.3) | 4.9 (0.1) | 5.1 (0.3)
Statistical Analysis 1: Comparison: Diet; Baseline vs 12 weeks. Statistical Analysis was performed only for the "Diet" Arm/Group; Test type: Superiority — Statistical Analysis was performed only for the "Diet" Arm/Group; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Body Composition
Description: Body Composition assessed by BMI
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 11 | 7 | 13 | 5
kg/m^2
  Baseline | 28.9 (2.5) | 30.8 (3.1) | 23.5 (2) | 29.1 (2)
  12 weeks | 28.6 (2.4) | 29.2 (3) | 23.5 (1.8) | 29.1 (2)
Statistical Analysis 1: Comparison: Diet; Baseline vs 12 weeks. Statistical Analysis was performed only for the "Diet" Arm/Group; Test type: Superiority — Statistical Analysis was performed only for the "Diet" Arm/Group; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Changes in Adipocyte Morphology
Description: Percentage Change in total adipose tissue assessed by MRI
Time Frame: 12 weeks
Population: 1 missing data in diet group
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 7 | 6 | 13 | 5
percentage change | -10.9 (5.1) | -8.9 (3.3) | -8.5 (2.7) | 3.7 (1.4)
Statistical Analysis 1: Comparison: Exercise; Baseline vs 12 weeks; Test type: Superiority; p < 0.05, t-test, 2 sided — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance
Statistical Analysis 2: Comparison: Diet; Baseline vs 12 weeks; Test type: Superiority; p < 0.05, t-test, 2 sided — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance
Statistical Analysis 3: Comparison: Exercise, Control; Baseline vs 12 weeks; Test type: Superiority; p < 0.05, t-test, 2 sided — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

5. Secondary Outcome: Genome Integrity (DNA Methylation and Telomere Length)
Time Frame: 12 weeks
Population: Data not collected
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Body Weight
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
Number analyzed (Participants) | 11 | 7 | 13 | 5
kg
  Baseline | 92.9 (9) | 91.9 (17.8) | 78.5 (2.3) | 84.7 (4.8)
  12 weeks | 91.6 (9.1) | 87.3 (17.4) | 78.3 (2.3) | 84.5 (4.9)
Statistical Analysis 1: Comparison: Diet; Baseline vs 12 weeks. Statistical Analysis was performed only for the "Diet" Arm/Group; Test type: Superiority — Statistical Analysis was performed only for the "Diet" Arm/Group; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Exercise | Diet | Exercise, Control | Diet, Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7 | 0/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/13 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes